CLINICAL TRIAL: NCT05674487
Title: Prostaglandins Versus Trans-Cervical Balloon for Induction of Labor in Fetal Growth Restriction: a Multicenter Open-label Randomized Trial
Brief Title: Prostaglandins Versus Trans-cervical Balloon for Induction of Labor in Fetal Growth Restriction (PROBIN)
Acronym: PROBIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: French Ministry of Social Affairs and Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2022/42; NCT05848869 (obsolete NCT alias)
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Fetal Growth Restriction
Keywords: Fetal growth restriction; Cesarean section; Induction of labor; Cervical ripening; Neonatal morbidity
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans-cervical balloon (Experimental): Induction of labor by cervical ripening with trans-cervical balloon (Foley catheter).
  Interventions: Device: Trans-cervical balloon
- Misoprostol (Active Comparator): Induction of labor by cervical ripening with Prostaglandins (Misoprostol per os)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Device: Trans-cervical balloon — Induction of labor by cervical ripening with trans-cervical balloon (Foley catheter).
  Arms: Trans-cervical balloon
Drug: Misoprostol — Induction of labor by cervical ripening with Prostaglandins (Misoprostol per os)
  Arms: Misoprostol

SUMMARY:
The goal of this randomized trial is to compare two methods of induction in a fetal growth restriction population. The main question it aims to answer is:

• Is trans-cervical balloon superior to prostaglandins in reducing the cesarean section rate, without increasing neonatal morbidity? Participants will have an induction of labour by cervical ripening with trans-cervical balloon in the trans-cervical balloon catheter arm and with Prostaglandins in the Misoprostol arm.

Researchers will compare two methods of induction: trans-cervical balloon and prostaglandins to see if trans-cervical balloon is associated with a lower risk of cesarean delivery.

DETAILED DESCRIPTION:
Fetal growth restriction (FGR) is associated with increased perinatal morbidity and mortality in late pregnancy. Because of this higher risk of adverse perinatal outcome, induction of labor is often proposed and require cervical ripening when the cervix is not favorable, i.e. Bishop score less than 6. Two methods of cervical ripening are currently available and used: pharmacological (prostaglandins) and mechanical (trans-cervical balloon).

Growth-restricted fetuses are a population at increased risk for non-reassuring fetal status and hypoxia during labor because of their lower weight. Prostaglandins can lead to cardiotocograph (CTG) tracing abnormalities by causing uterine tachysystole in normal-weight fetuses. Nevertheless, the question of the method of induction of labor has been poorly studied in the population of growth-restricted fetuses. None of the national and international societies reports in their guidelines which method of induction of labor should be offered to pregnancies complicated by a fetal growth restriction. A few retrospective studies are in favor of an increased risk of uterine tachysystole with consequences on the CTG tracing in the case of cervical ripening with prostaglandins compared to the trans-cervical balloon. However, the results of these studies lack robustness due to important methodological limitations.

Because trans-cervical balloon is a mechanical method of cervical ripening, it may be less likely to cause uterine tachysystole and thus fewer non-reassuring fetal status. Thus, the risk of cesarean section in labor could be decreased compared with the use of prostaglandins in the growth-restricted fetal population.

To date, there is no published quality randomized controlled trials on the optimal method of cervical ripening in induction of labor for FGR fetuses.

The present large-scale randomized trial aim to define the preferred method of induction for these fetuses, associated with a lower risk of cesarean delivery. If it is demonstrated that one method of induction (trans-cervical balloon) is superior to another (prostaglandins) in reducing the cesarean section rate, without increasing neonatal morbidity, the results of our study are likely to lead to changes in national and international recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Singleton gestation, with cephalic presentation
* Gestational age at randomization between entre 34 weeks of gestation and 0 day and 41 weeks of gestation and 0 day
* Fetal growth restriction (FGR). FGR is defined at the third trimester by an abdominal circumference below the 10th centile and/or an estimated fetal weight below the 10th centile (according to local curve), according to the trial DIGITAT. Fetus with normal and abnormal Doppler index can be included.
* Plan for induction of labor whatever the indication (fetal growth restriction or other), the induction of labor is the induction of birth by vaginal delivery
* Bishop Score below 6
* Affiliated or beneficiary to a health security system
* Signed informed consent

Exclusion Criteria:

* Contraindication to an induction of labor
* History of previous cesarean delivery, myomectomy by laparotomy or laparoscopy
* Contraindication to misoprostol or trans-cervical balloon
* Known HIV positivity (because of modified delivery plan)
* Known major fetal anomaly or chromosomic anomaly
* Fetal demise
* Patient under legal protection
* Poor understanding of the French language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 774 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
cesarean section | Day 1
  Incidence of cesarean section defined as a cesarean birth regardless of the indication

SECONDARY OUTCOMES:
duration of labor | Day 1
  Mean duration of labor (duration between admission to the labor room and delivery)
duration between cervical ripening and delivery | Day 1
  Mean duration between cervical ripening and delivery
oxytocin use | Day 1
  Incidence of oxytocin use (median of the maximal administered dosage)
operative delivery | Day 1
  Incidence of operative delivery (vacuum, forceps, spatula)
postpartum hemorrhage | Day 3
  Incidence of postpartum hemorrhage defined by blood loss >500mL (defined according to the CNGOF criteria)
Mean total blood loss | Day 3
  Mean total blood loss (mL)
intra-uterine infectious | Day 5
  Incidence of intra-uterine infectious defined by a fever (maternal temperature equal to or greater than 38°C twice), associated to at least one of the two criterion: persistent fetal tachycardia > 160 bpm, or purulent amniotic fluid (defined according to the CNGOF criteria).
iron administration | Day 5
  Incidence of postpartum intravenous iron administration
transfusion | Day 5
  Incidence of transfusion of blood products or blood
maternal thromboembolism event | Day 5
  Incidence of maternal thromboembolism event (deep venous thrombosis diagnosed using leg Doppler ultrasound or pulmonary embolism diagnosed using computed tomographic pulmonary angiography)
maternal satisfaction | Day 5
  Incidence of maternal satisfaction with a satisfaction questionnaire derived from the childbirth experience questionnaire and satisfaction questionnaire of TRAAP2 study
Mean duration of hospitalization | Day 5
  Mean duration of hospitalization
umbilical artery lactic acid | Day 1
  Incidence of umbilical artery lactic acid greater than 10mmol/l
umbilical artery pH | Day 1
  Incidence of umbilical artery pH of less than 7,05
neonatal Apgar Score | Day 1
  Incidence of neonatal 5 minutes Apgar Score of less than 7
neonatal hypoglycemia | Day 5
  Incidence of neonatal hypoglycemia (blood glucose < 35 mg/L) requiring intravenous therapy
neonatal intensive care | Day 5
  Incidence of admission to neonatal intensive care unit or intermediate care unit
neonatal length of hospital stay | Day 5 up to Month 2
  Mean neonatal length of hospital stay
neonatal death before discharge | Day 1 up to Month 2
  Incidence of neonatal death before discharge
non-reassuring fetal status | Day 1
  Incidence of non-reassuring fetal status occurring after the beginning of the cervical ripening (including both cervical ripening and labor). Non-reassuring fetal status is defined by the Fédération Internationale de Gynécologie et d'Obstétrique (FIGO), who class the CTG tracing in 3 class: normal, suspicious and pathological 3. According to this classification, non-reassuring fetal status is defined as the presence of a suspicious or pathological CTG tracings, predictive of hypoxia/ neonatal acidosis status
cesarean section for non-reassuring fetal status | Day 1
  Incidence of cesarean section for non-reassuring fetal status
cesarean section for arrest of labor | Day 1
  Incidence of cesarean section for arrest of labor
neonatal ventilation | Day 3
  Incidence of the need for neonatal ventilation in the first 72 hours of life, defined by intubation, continuous positive airway pressure (CPAP) or high-flow nasal cannula
neonatal hypoxic-ischemic encephalopathy | Day 1 up to Month 2
  Incidence of neonatal hypoxic-ischemic encephalopathy
neonatal seizure | Day 1
  Incidence of neonatal seizure
neonatal infection | Day 1 up to Day 28
  Incidence of neonatal infection (confirmed sepsis or pneumonia)
neonatal meconium aspiration syndrome | Day 5
  Incidence of neonatal meconium aspiration syndrome,
birth trauma | Day 5
  Incidence of birth trauma (bone fracture, neurologic injury, or retinal hemorrhage),
neonatal intracranial or subgaleal hemorrhage | Day 5
  Incidence of neonatal intracranial or subgaleal hemorrhage,
neonatal arterial hypotensio | day 1
  Incidence of neonatal arterial hypotension requiring pressor support
Maternal Postpartum Depression | 2 months after delivery.
  Defined by a score greater than 13 on the EPDS (Edinburgh Postpartum Depression Scale). The EPDS scale calculates a depressive symptom score ranging from 0 (no depression symptoms) to 30 (severe depression symptoms). Threshold values greater than 13 are used to identify women at high risk for postpartum depression.
Posttraumatic Stress Disorder (PTSD) | 2 months after delivery.
  Defined by a score greater than 33 on the IES-R (Impact of Event Scale - Revised) questionnaire or by the presence of all criteria from the DSM-IV (4th edition of the Diagnostic and Statistical Manual of Mental Disorders) (criteria A, B, C, D, E, and F) on the TES (Traumatic Event Scale). The IES-R measures the severity of PTSD symptoms over the past 7 days, with scores ranging from 0 (no PTSD symptoms) to 88 (extreme PTSD symptoms). The diagnosis of PTSD is made when the IES-R score is greater than 33.
  • Timeframe:

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No